CLINICAL TRIAL: NCT03171298
Title: Laparoscopic Assisted Transanal Resection of Rectal Cancer With Total Mesorectal Excision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed abulfetouh, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: transanal surgical approach
Record Dates: First submitted 2017-05-20; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transanal TME (Experimental): Laparoscopic Assisted Transanal Total Mesorectal Excision
  Interventions: Procedure: Laparoscopic Assisted Transanal Total Mesorectal Excision

INTERVENTIONS:
Procedure: Laparoscopic Assisted Transanal Total Mesorectal Excision — * Abdominal approach with laparoscopic mobilization of the left colon
  * Laparoscopic isolation and transection of inferior mesenteric vessels .
  * Transabdominal dissection of the upper rectum and mesorectam.
  * Insertion of transanal platform and the creation of pneumorectum.
  * Occlusion of rectum 2 cm distal to the rectal lesion via purse string.
  * Transanal dissection of lower and mid mesorectam
  * The specimen will be extracted transanally

SUMMARY:
Rectal cancer is one of the frequent malignant neoplasms ,Total mesorectal excision (TME) has become the gold standard treatment for middle and lower rectal cancers. Laparoscopic TME still be difficult in patients with low rectal tumors, narrow pelvic anatomy, male sex or high body mass index . Difficult visualization of the pelvic anatomy along with the limitation of rigid laparoscopic instruments may affect the quality of oncological outcomes and increase the risks of injuries during surgery. A down to up approach via transanal total mesorectal excision (TaTME) technique may overcome these problems

DETAILED DESCRIPTION:
This clinical trial will be conducted at general surgery department of Assiut University Hospital .

.

ELIGIBILITY:
Inclusion Criteria:

* • rectal cancer histologically proven through biopsy

  * tumours located at least 3 cm from anorectal ring;
  * local spread restricted to the rectal wall
  * adequate preoperative sphincter function and continence;
  * absence of distant metastases.
  * Suitable for elective surgical resection

Exclusion Criteria:

* • T4 tumours not responding to neoadjuvant chemo- radiotherapy

  * Patients under 18 years of age
  * Pregnancy
  * Previous rectal surgery (except local excision, endoscopic mucosal resection (EMR) or polypectomy)
  * Patients with acute intestinal obstruction
  * Multiple colorectal tumours
  * Familial Adenomatosis Polyposis Coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), Crohn's disease or ulcerative colitis
  * Planned synchronous abdominal organ resections
  * Preoperative evidence for distant metastases through imaging of the thorax and abdomen
  * Absolute contraindications to general anaesthesia,
  * presence of fecal incontinence,
  * undifferentiated tumors .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
intraoperative complication | 1 day
  complication occured intraoperatively or on the first day of surgery

SECONDARY OUTCOMES:
resection margin | 1 years
  circumferential resection margin microscopic examination
Mortality rate | 1 years
  rate of death
morbidity rate | 1 year
  rate of postoperative morbidity
recurrance rate | 2 years
  rate of local recurance( by CT scan )
Anorectal function outcomes | 2 years
  manometric assessment of anorectal function
Sexual functional outcomes | 2 years
  sexual function with IIEF(International Index of Erectile Function) questionnaire
Mesorectal completeness | 1 year
  The quality of the mesorectum or TME specimen(pathological examination)

CONTACTS AND LOCATIONS:
Overall Officials: samir a ali, phd, Study Director — assuit university hospital
Locations (1):
- Assuit Universty Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang L, Chen WH, Luo SL, Luo YX, Liu ZH, Huang MJ, Wang JP. Transanal total mesorectal excision for rectal cancer: a preliminary report. Surg Endosc. 2016 Jun;30(6):2552-62. doi: 10.1007/s00464-015-4521-2. Epub 2015 Aug 27. PMID 26310534